CLINICAL TRIAL: NCT01200134
Title: Hypoxia Diagnosis and Evaluation Using F-MISO PET and Biomarkers in Brain Tumors
Brief Title: HYPONCO - Hypoxia in Brain Tumors
Acronym: HYPONCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-015543-16
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Anaplastic Glioma
Keywords: glioma patients : anaplasic glioma (grade III) and GBM (grade IV)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FMISO PET-scanning (Experimental): Other: 18F-FMISO PET-scanning 18F-FMISO PET-scanning: 18F-FMISO PET-scanning will be performed at the same place following the same protocol as mentioned above. However, the 20-minutes period of PET images acquisition will start 120 minutes after the 18F-FMISO bolus injection (0.05 mCi/kg).
  Interventions: Other: 18F-FMISO PET-scanning

INTERVENTIONS:
Other: 18F-FMISO PET-scanning — Other: 18F-FMISO PET-scanning 18F-FMISO PET-scanning: 18F-FMISO PET-scanning will be performed at the same place following the same protocol as mentioned above. However, the 20-minutes period of PET images acquisition will start 120 minutes after the 18F-FMISO bolus injection (0.05 mCi/kg).

SUMMARY:
Background :

In malignant gliomas, hypoxia is associated with tumour angiogenesis and tumour progression. This multidisciplinary preclinical and clinical project aims to validate the use of 18F-FMISO as a hypoxic marker for diagnosis, treatment and follow-up of malignant gliomas. Indeed, non-invasive methods of imagery such as Positron Emission Tomography (PET) and biological methods (after surgical resection) to detect the endogenous expression of factors induced by the hypoxia would allow to identify hypoxic areas. Identifying, with accuracy, the hypoxic areas could allow the clinicians to evaluate the response to the anti-angiogenic agents (preliminary validation in the preclinical project) and to optimize the combination of the anti-VEGF treatments with other conventional therapeutic approaches (radiotherapy, chemotherapy or other molecules).

Research project :

This research project includes 3 steps : first the investigators will establish the 18F-FMISO production technique for clinical application at CYCERON PET center. The second step consists in the preclinical validation of 18F-FMISO as a hypoxic marker and as a powerful tool for evaluating the therapeutical efficiency of anti-angiogenic treatment (sutent) in experimental rat gliomas. The third step is the clinical trial HypOnco. This research proposal aims to develop and use non invasive imaging methods (18F-FMISO with PET) and biological methods (after surgical resection) to detect hypoxic (HIF1 and HIF2) and angiogenic (VEGF and EPO) regions in different malignant gliomas with different degrees of vascularization (15 patients with grade III gliomas and 15 patients with grade IV glioblastomas). Within the same patient 18F-FMISO as a hypoxic index will be performed. A magnetic resonance imaging examination (MRI) including perfusion sequences and MR spectroscopy will also be assessed for each patient. Following this imaging protocol, surgical resection will be performed allowing us to study expression of endogenous factors induced by hypoxia and angiogenic factors by real time RT-PCR and in immunohistochemistry.

The data obtained will enable us to establish :

* a hypoxic index (18F-FMISO with PET).
* an index of hypoxic factor expression (HIFs)
* an angiogenic index (VEGF, EPO, vascular markers)

The investigators will characterize the links between these data and also with the following parameters:

* clinical (age, Karnofsky performance status, survival)
* MR parameters included perfusion and spectroscopy
* histological (necrosis, cellular proliferation, atypical cell abnormalities, vascularization).

Expected results and clinical advantages

* To establish the 18F-FMISO production technique
* To propose the 18F-FMISO as a non-invasive marker for efficacy of antiangiogenic treatment in a preclinical study.
* To define the relationship between the 18F-FMISO uptake and tumour grade, patient survival, tumour recurrence, expression of hypoxic and angiogenic factors and tumour vascularisation.
* To provide a hypoxic index in cerebral tumours from 18F-FMISO PET, allowing diagnosis and prognosis improvement for optimal treatment orientation and strategy.

In the field of the clinical applications, this tool will allow to :

* Optimize radiotherapy treatment by identifying with accuracy, using 18F-FMISO PET, the most hypoxic areas which are also the most radio resistant.
* Evaluate antiangiogenic therapy efficacy

ELIGIBILITY:
Inclusion Criteria:

* adults aged >= 18 years
* KPS >= 70%
* must have the understanding and ability to sign an informed consent document
* be male or non-pregnant
* non-lactating females
* Patients who are fertile must agree to use an effective method of contraception during participation in the study
* the following laboratory results : absolute neutrophil count >= 1500 cells/µl, platelet count >= 100,000 cells/µl, SGOT <= 2.5 x ULN, serum creatinine <= 1.5 x ULN

Exclusion Criteria:

* contraindication to surgery
* concomitant radio-, chemo-, or immunotherapy
* known diagnosis of Human Immunodeficiency Virus (HIV) infection
* patient with hepatitis B or C
* diabetic patient
* patient with kidney or liver deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
hypoxia volume (HV) and degree (maximum ratio [Rmax]) defined from 18F-FMISO uptake rates | PET 18F-MISO between Day 1 & Day 7
  * determine, in vivo, the hypoxic character of tumours from a PET biomarker. Tumoral hypoxia will be characterized by hypoxia volume (HV) and degree (maximum ratio [Rmax]) defined from 18F-FMISO uptake rates
  * characterize the link between the tumoral hypoxia and the hypoxic and angiogenic factor expressions that favour vascular neoformation and proliferation feeding tumoral cells

CONTACTS AND LOCATIONS:
Overall Officials: GUILLAMO Jean Sébastien, MD, PhD, Principal Investigator — University Hospital, Caen; DERLON Jean Michel, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France